CLINICAL TRIAL: NCT02986633
Title: Prediction of Response to Cardiac Resynchronization Therapy by New Echocardiographic Methods
Brief Title: Echocardiography in Cardiac Resynchronization Therapy (Echo-CRT)
Acronym: Echo-CRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-009
Record Dates: First submitted 2016-12-05; First posted 2016-12-08 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: Cardiac Resynchronization Therapy; Echocardiography; Biventricular Pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with heart failure and CRT: Heart failure with left ventricular ejection fraction less than 35 % treated with CRT
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography

SUMMARY:
The present observational prospective study aims at identifying echocardiographic parameters (based on the Left Bundle Branch Block (LBBB)-like contraction of the left ventricle (LV) ascertained using new methods of echocardiography including speckle tracking strain) that are linked to Cardiac Resynchronization Therapy (CRT) response and a better outcome following CRT

DETAILED DESCRIPTION:
The Cardiac Resynchronization Therapy (CRT) reduces mortality of patients with heart failure and reduced LV ejection fraction. The clinical benefit of CRT is mediated by LV reverse remodelling (decrease in LV end-systolic volume over time). However, 30 to 50 % of these patients will not experience LV reverse remodelling following CRT.

Classical parameters of dyssynchrony obtained by conventional methods of echocardiography (including doppler tissue imaging) have a limited value in predicting CRT response. Meanwhile, patients with a Left Bundle Branch Block (LBBB) on the electrocardiogram experience more frequently LV reverse remodelling than those without a LBBB.

LBBB is responsible for specific LV contractile abnormalities that can be identified by speckle tracking strain echocardiography (early septal contraction, stretching of late contraction of the postero-lateral wall). The predictive value of these abnormalities remains to be studied.

Thus, it has been hypothesised that these LBBB-related contractile abnormalities may be independent predictors of LV reverse remodelling and outcome following CRT.

The present observational prospective study aims at identifying echocardiographic parameters (based on the LBBB-like contraction of the LV ascertained using new methods of echocardiography including speckle tracking strain) that are linked to CRT response and a better outcome following CRT.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with left ventricular ejection fraction less than 35 %
* QRS duration over than 120 ms
* Clinical indication for CRT

Exclusion Criteria:

* Rythmologic indication of CRT for atrial fibrillation control
* Rythmologic indication of CRT for left ventricular ejection fraction between 35% and 45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with LV systolic dysfunction and QRS duration > 120 ms receiving CRT at GHICL.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-12; Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in left ventricular end-systolic volume measured by echocardiography | 9 months after implantation

SECONDARY OUTCOMES:
Death rate | 2, 4, 6, 8 and 10 years after implantation
re-hospitalisation rate | 2, 4, 6, 8 and 10 years after implantation
Changes in left ventricular ejection fraction measured by echocardiography | 9 months after implantation
Changes in left ventricular end-diastolic volume measured by echocardiography | 9 months after implantation
Changes in left ventricular longitudinal strain measured by echocardiography | 9 months after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Sylvestre Maréchaux, MD, PhD, Principal Investigator — Hospital of Lille Catholic University (GHICL)
Locations (1):
- Hospitals of Lille Catholic University (GHICL), Lomme, France

REFERENCES:
- [Derived] Layec J, Decroocq M, Delelis F, Appert L, Guyomar Y, Riolet C, Dumortier H, Mailliet A, Tribouilloy C, Marechaux S, Menet A. Dyssynchrony and Response to Cardiac Resynchronization Therapy in Heart Failure Patients With Unfavorable Electrical Characteristics. JACC Cardiovasc Imaging. 2023 Jul;16(7):873-884. doi: 10.1016/j.jcmg.2022.12.023. Epub 2023 Mar 8. PMID 37038875
- [Derived] Appert L, Menet A, Altes A, Ennezat PV, Bardet-Bouchery H, Binda C, Guyomar Y, Delelis F, Castel AL, Le Goffic C, Guerbaai RA, Graux P, Tribouilloy C, Marechaux S. Clinical Significance of Electromechanical Dyssynchrony and QRS Narrowing in Patients With Heart Failure Receiving Cardiac Resynchronization Therapy. Can J Cardiol. 2019 Jan;35(1):27-34. doi: 10.1016/j.cjca.2018.10.019. Epub 2018 Nov 14. PMID 30595180